CLINICAL TRIAL: NCT00509223
Title: Effect of PAP Treatment on Glycemic Control in Patients With Type 2 Diabetes and Obstructive Sleep Apnea
Brief Title: GLYCOSA Study:Effect of PAP Treatment on Glycemic Control in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: Royal North Shore Hospital (Other); Baker Heart and Diabetes Institute (Other); International Diabetes Center at Park Nicollet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA-09-06-01
Record Dates: First submitted 2007-07-29; First posted 2007-07-31 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Type 2 diabetes; Obstructive sleep apnea; Glycemic control; Insulin resistance; Sleep disordered breathing
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Apnea, Obstructive; Insulin Resistance; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Lifestyle counseling with Positive Airway Pressure (PAP) therapy
  Interventions: Device: Positive Airway Pressure therapy; Behavioral: Lifestyle counseling
- Group 2 (Active Comparator): Lifestyle counseling without Positive Airway Pressure (PAP) therapy
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Device: Positive Airway Pressure therapy — Positive Airway Pressure (PAP) therapy initiated at Randomization and continued through the entire study duration (6 months), with instructions for use on a daily basis, during periods of sleep.
  Other Names: ResMed AutoSet S8
  Arms: Group 1
Behavioral: Lifestyle counseling — Lifestyle counseling: All subjects were counseled regarding adopting a healthy lifestyle and advised on the Heart Foundation, National Health and Medical Research Council, and American Diabetes Association nutrition and exercise recommendations.

SUMMARY:
Obstructive Sleep Apnea (OSA) and type 2 diabetes mellitus are two prevalent medical conditions with significant associated cardiovascular and cerebrovascular morbidity and mortality. Research indicates that the prevalence of OSA is increased in diabetic patients when compared with normoglycemic patients and that OSA is independently associated with type 2 diabetes. Further research suggests that effective treatment of the OSA with continuous positive airway pressure (CPAP) improves insulin responsiveness in both non-diabetic OSA patients and diabetic-OSA patients. We are proposing a clinical trial to evaluate the impact of 6 months of CPAP therapy on glycemic control in type 2 diabetic patients with OSA.

The primary objective of this study is to assess the effectiveness of CPAP in improving glycemic control (HbA1c) in type 2 diabetic patients with newly diagnosed OSA. Secondary objectives of this study include: assessment of fasting and post prandial glucose, determination as to whether there are any biochemical markers for OSA in the type 2 diabetic population; assessment of any improvements in cardiovascular outcomes; evaluation of any improvement in quality of life. Patients with OSA will be randomized into one of two groups: either a CPAP treatment group or a non-treatment group. Patients will be followed at 3 months and 6 months with collection of various lab tests to assess glycemic control.

DETAILED DESCRIPTION:
Patients attending clinical sites involved with the trial will be asked to participate in the study. Patients will undergo a sleep test and if positive for Obstructive Sleep Apnea (OSA) will continue in the study.

At the time of enrolment baseline history and physical examination will be assessed. Baseline lab samples will also be obtained to measure levels of fasting blood glucose, insulin, HbA1c, lipids, biochemical markers and creatinine/albumin ratio. Post-prandial glucose levels and 24-hour ambulatory blood pressure will be evaluated. Participants will also be asked to complete Quality of Life (QoL) questionnaires.

Participants will be randomised into either continuous positive airway pressure CPAP treatment or no treatment. All subjects will be counselled regarding adopting a healthy lifestyle and advised on the Heart Foundation, National Health and Medical Research Council, and American Diabetes Association nutrition and exercise recommendations. Follow-up on adoption of the healthy lifestyle approach will be done for all study participants for the duration of the trial period. Total duration of a patient's participation is 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older,
2. Known diagnosis of type 2 diabetes for at least 3 months
3. HbA1c >6.5% and </= 8.5%
4. BMI </= 40 kg/m2

Exclusion Criteria:

1. Requires oxygen therapy
2. OSA is severe (AHI>70 or SaO2<70%)
3. Work in transport related industries
4. Previous diagnosis of OSA
5. Known MVA due to sleepiness in the previous 5 years
6. Insulin-requiring
7. Use of GLP-1 mimetic (e.g. Byetta) for < 6 months or > 6 months but weight not stable
8. Unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2007-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Zimmet, MBBS MD PhD, Study Chair — International Diabetes Institute, Australia
Locations (15):
- United States (11):
  - Mission Internal Medical Group, Mission Viejo, California
  - Advanced Metabolic Care and Research Institute, Temecula, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - SleepMed of Central Georgia, Macon, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - International Diabetes Center, Saint Louis Park, Minnesota
  - Rochester Clinical Research, Rochester, New York
  - OSU Sleep Medicine Program, Columbus, Ohio
  - SleepMed of West Ashley, Charleston, South Carolina
  - SleepMed of South Carolina, Columbia, South Carolina
  - Cetero Research, San Antonio, Texas
- Australia (3):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Baker IDI Heart and Diabetes Institute, Melbourne, Victoria
- IUCPQ, Québec, Quebec, Canada

REFERENCES:
- [Derived] Shaw JE, Punjabi NM, Naughton MT, Willes L, Bergenstal RM, Cistulli PA, Fulcher GR, Richards GN, Zimmet PZ. The Effect of Treatment of Obstructive Sleep Apnea on Glycemic Control in Type 2 Diabetes. Am J Respir Crit Care Med. 2016 Aug 15;194(4):486-92. doi: 10.1164/rccm.201511-2260OC. PMID 26926656

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for this study were recruited from 15 medical clinics located in the United States and Australia.
Pre-assignment Details: Subjects were presented with an Informed Consent Form (and HIPAA in USA) and assessed for eligibility based on inclusion /exclusion criteria. If all IEC met, subjects randomized 1:1. 118 subjects not included in endpoint analysis due to reanalysis of Obstructive Sleep Apnea (OSA) inclusion criteria. 298 of the 416 were included for final analysis.
Groups:
- Group 1: Lifestyle counseling with Positive Airway Pressure (PAP) therapy
  Lifestyle counseling: All subjects were counseled regarding adopting a healthy lifestyle and advised on the Heart Foundation, National Health and Medical Research Council, and American Diabetes Association nutrition and exercise recommendations.
  Positive Airway Pressure therapy : PAP therapy was initiated at Randomization and continued through the entire study duration (6 months), with instructions for use on a daily basis, during periods of sleep.
- Group 2: Lifestyle counseling without Positive Airway Pressure (PAP) therapy
  Lifestyle counseling: All subjects were counseled regarding adopting a healthy lifestyle and advised on the Heart Foundation, National Health and Medical Research Council, and American Diabetes Association nutrition and exercise recommendations.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 207 | 209
Completed | 119 | 137
Not Completed | 88 | 72
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 25 | 6
Not completed — Including: subject change of address | 5 | 2
Not completed — Did not meet revised inclusion criteria | 56 | 62

BASELINE CHARACTERISTICS:
Population: 118 subjects (of the 416 that started in the participant flow module) were not included in endpoint analysis due to reanalysis of OSA inclusion criteria. Thus, 298 of the 416 were included for final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling With PAP Therapy | Lifestyle Counseling | Total
Number analyzed (Participants) | 151 | 147 | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 90 | 174
  >=65 years | 67 | 57 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (9.1) | 62.1 (9.0) | 62.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 106
  Male | 99 | 93 | 192
Region of Enrollment [Number; unit: participants]
  United States | 54 | 59 | 113
  Australia | 97 | 88 | 185

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change
Description: Month 6 change in HbA1c (%)
Time Frame: Baseline to Month 6
Population: The following definition was applied to the primary endpoint: included in analysis were all participants that had at least 1 follow-up HbA1c value in addition to the Baseline HbA1c were considered.
Measure: Mean (Standard Deviation); unit: HbA1c percent
Arm/Group | Lifestyle Counseling With PAP Therapy | Lifestyle Counseling
Number analyzed (Participants) | 129 | 138
HbA1c percent | -0.1 (0.8) | -0.1 (0.7)

ADVERSE EVENTS:
Arm/Group | Lifestyle Counseling | Lifestyle Counseling With PAP Therapy
Serious Adverse Events (participants affected / at risk) | 5/147 | 10/151
Other Adverse Events (participants affected / at risk) | 78/147 | 94/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Counseling (N=147) | Lifestyle Counseling With PAP Therapy (N=151)
GI Distress (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Procedure (Surgical and medical procedures) | 2 (2) | 2 (2)
TIA / Blockage of Artery (Cardiac disorders) | 0 (0) | 2 (2)
Ovarian Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Brachial Plexopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lifestyle Counseling (N=147) | Lifestyle Counseling With PAP Therapy (N=151)
GI Distress (Gastrointestinal disorders) | 5 | 9
General Infection (Blood and lymphatic system disorders) | 8 | 6
Nasal Dryness/Irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Pain (Musculoskeletal and connective tissue disorders) | 17 | 11
Skin Irritation (Skin and subcutaneous tissue disorders) | 11 | 19
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 34 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less